CLINICAL TRIAL: NCT07126613
Title: Development of a Just-in-Time Adaptive Intervention to Reduce High-Intensity Drinking Among Young Adults
Brief Title: Mobile Alcohol Use Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25-1872; K01AA028540 (NIH)
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Misuse
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Health Intervention (Experimental): Participants will receive access to the mobile health intervention. This includes access to an online dashboard which includes a drink counter, ability to track the number of drinks consumed over the course of the study, ability to set drinking-related goals for oneself, and alcohol-related resources. Participants in the intervention will also receive tailored messages during drinking episodes which target contextual factors to reduce alcohol use.
  Interventions: Behavioral: Mobile Health Intervention to Reduce Alcohol Use Among Young Adults
- No-contact control (No Intervention): Participants will receive only morning surveys and the 30-day post-test survey.

INTERVENTIONS:
Behavioral: Mobile Health Intervention to Reduce Alcohol Use Among Young Adults — The mobile just-in-time adaptive intervention consists of 1) a digital participant dashboard and 2) tailored messages delivered to the participant's cellphone addressing the individual and ecological contexts of alcohol use.
  The web-based intervention dashboard includes: 1) a drink counter for participants to log the number and type of drinks (e.g., beer, wine, mixed drink) they consume in a drinking occasion; 2) a calendar which summarizes the number of days on which a participant has consumed alcohol and the number of drinks consumed over the study period, broken out by drink type; 3) a log where participants can set drinking-related goals and update their progress on those goals; and 4) national and local substance use resources.
  Participants will receive messages tailored to their drinking situation and ecological context during high-risk drinking times.
  Arms: Mobile Health Intervention

SUMMARY:
This study aims to examine the feasibility and acceptability of a mobile health intervention to reduce alcohol use and related consequences among young adults. Participants will be randomly assigned to either receive access to the mobile health intervention or receive only generic study surveys. Participants will receive text message surveys sent to their personal cellphone for 4 weeks per their assigned trial arm. All participants will receive a post-survey 30 days after their final weekly survey text.

DETAILED DESCRIPTION:
This study aims to determine whether a mobile health intervention to reduce alcohol use and related consequences is acceptable and feasible among young adults who engage in high-intensity drinking (HID; 8+/10+ drinks per drinking occasion for females/males, respectively). The investigators aim to recruit 40 adults between 18-25 years of age who report at least one HID episode in the past 30 days.

After providing informed consent, participants will be randomly assigned to receive the mobile health intervention or control surveys only.

Participants will attend one online study visit to enroll in the study and be assigned to their study arm. All subsequent study activities will be completed asynchronously. Participants will then receive text message prompts and/or surveys to their personal cellphone either Wednesday or Thursday through Sunday for four consecutive weeks. Participants will receive a post-test survey 30 days after their final weekly survey.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25
* Experience at least one high-intensity drinking episode in the past 30 days
* Able to read and write in English
* Consent to receiving text messages to personal cellphone
* No current history of substance use treatment in the past 12 months
* Did not participate in the Aim 2 technical field trial of the intervention

Exclusion Criteria:

* Under 18 or over 25
* Did not experience at least one high-intensity drinking episode in the past 30 days
* Unable to read and write in English
* Does not consent to receive text messages to personal cellphone
* Current or history of substance use treatment in the past 12 months
* Participated in the Aim 2 technical field trial of the intervention

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-01-06 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
Average Satisfaction with the Intervention | Assessed 30 days after the last 4-week survey text.
  Measured using the following item, "How satisfied are you with your experience using this intervention?" with a 5-point response scale ranging from Not at All Satisfied (1) to Extremely Satisfied (5). A higher score indicates higher satisfaction with the intervention
Average Engagement with the Intervention Measured by the DCBI Scale | Assessed 30 days after the last 4-week survey text.
  Engagement will be assessed via 8 items from the Digital Behavior Change Intervention (DCBI) Scale. The item stem "How strongly did you experience the following?" will be repeated for the following concepts: interest, intrigue, focus, inattention, distraction, enjoyment, annoyance, and pleasure. All items will be scored on a 7 point scale from Not at All (1) to Extremely (7) and an average composite score will be derived for each participant based on responses across the seven items. Scores range from 1-7, where a higher score indicates higher engagement with the intervention.

SECONDARY OUTCOMES:
Number of Drinks Consumed per Drinking Episode | Four days per week (Thursday-Sunday) for four consecutive weeks (16 total times).
  Total number of drinks consumed per drinking occasion will be assessed using 1 item: "How many standard drinks did you consume yesterday?" Response options will range from less than 1 (0) to 10 or more (10). Respondents who input 10 or more drinks will be prompted to input the total number of drinks they consumed.
Average Drinking Level per Drinking Episode | Four days per week (Thursday-Sunday) for four consecutive weeks (16 total times).
  An ordinal measure of drinking level will be calculated based on the total drinks item ("How many standard drinks did you consume yesterday?"). Moderate drinking will be defined as 0-3 drinks for women or 0-4 drinks for men, standard binge drinking will be defined as 4-7 drinks for women or 5-9 drinks for men, and high-intensity drinking will be defined as 8 or more drinks for women or 10 or more drinks for men.
Frequency Score of Alcohol-Related Consequences Measured by BYAACQ | Assessed 30 days after the last 4-week survey text.
  Alcohol-related consequences will be measured via the 24-item Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ), which lists a variety of alcohol-related consequences and asks participants to endorse (Yes=1; No=0) if they have experienced a specific consequence in the past month. Scores range from 0-24, where a higher score indicates a higher number of alcohol-related consequences experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa J Cox, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Rosenau Hall, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigator will post de-identified participant data to the National Institute of Mental Health National Data Archive (NDA).
Time Frame: Data will become available 9/1/2027 and be hosted indefinitely on the NDA repository.
Access Criteria: Individuals who meet the data access eligibility criteria set by the NDA may access the IPD.

DOCUMENTS (1):
  • Informed Consent Form (2025-09-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT07126613/ICF_000.pdf